CLINICAL TRIAL: NCT01887002
Title: A Phase 2, Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled Study to Evaluate the Effects of ONO-2952 on Pain Perception Produced by Rectal Distention in Female Subjects With Diarrhea-Predominant Irritable Bowel Syndrome (IBS-D) (RESTORE)
Brief Title: Study to Evaluate the Effects of ONO-2952 on Pain Perception Produced by Rectal Distention in Female Subjects With Diarrhea-Predominant Irritable Bowel Syndrome (IBS-D)
Acronym: RESTORE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to slow accrual of subjects.
Sponsor: Ono Pharma USA Inc (Industry)
Responsible Party: Sponsor
Organization: Ono Pharmaceutical Co. Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-2952POU005
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-01

CONDITIONS: Irritable Bowel Syndrome (IBS)
Keywords: Irritable Bowel Syndrome; IBS; ONO-2952
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — ONO-2952

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Arm 1 (Experimental): ONO-2952 Active tablets, every day for 2 weeks
  Interventions: Drug: ONO-2952
- Placebo Arm (Placebo Comparator): ONO-2952 Matching Placebo every day for 2 weeks
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: ONO-2952 — ONO-2952 Active tablets, every day for 2 weeks
  Arms: Experimental Arm 1
Drug: Placebo comparator — ONO-2952 Matching Placebo every day for 2 weeks
  Arms: Placebo Arm

SUMMARY:
The objective is to evaluate whether ONO-2952 modulates visceral pain perception produced by rectal distention in female patients with IBS-D

ELIGIBILITY:
Inclusion Criteria:

1. Female 18-65 years of age (inclusive)
2. Diagnosed with IBS based on the following criteria (Rome III criteria):

   * Symptom onset at least 6 months prior to diagnosis, and
   * Recurrent abdominal pain or discomfort at least 3 days per month for the past 3 months, and
   * Abdominal discomfort or pain associated with two or more of the following at least 25% of the time:
   * improvement with defecation
   * onset associated with a change in frequency of stool/defecation
   * onset associated with a change in form (appearance) of stool
3. Diagnosed with IBS-D, defined as loose/watery stools ≥ 25% and hard/lumpy stools ≤ 25% of defecations

Exclusion Criteria:

* Any structural abnormality of the gastrointestinal (GI) tract (other than esophagitis or gastritis)
* History of Chron's disease, ulcerative colitis, diabetes mellitus, lactose malabsorption, malabsorption syndromes, celiac sprue, or any upper GI symptoms that may impact the assessment of IBS symptoms

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-06; Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity rating during rectal distention by using a numeric pain rating scale | 2 weeks

SECONDARY OUTCOMES:
Safety assessed through adverse events and clinical laboratory values | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ono Pharma USA, Inc., Study Director — Ono Pharmaceutical Co. Ltd
Locations (4):
- United States (4):
  - Boston Clinical Site, Boston, Massachusetts
  - St. Louis Clinical Site, St Louis, Missouri
  - Chapel Hill Clinical Site, Chapel Hill, North Carolina
  - Oklahoma City Clinical Site, Oklahoma City, Oklahoma